CLINICAL TRIAL: NCT04612868
Title: Pivotal Prospective Clinical Trial to Demonstrate the Efficacy and Safety of AEYE-DS Software Device for Automated Diabetic Retinopathy Detection From Digital Fundoscopic Images
Brief Title: Efficacy and Safety of AEYE-DS Software Device for Automated Detection of Diabetic Retinopathy From Digital Fundus Images
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AEYE Health Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AEYE-DS-001
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AEYE Software Device (Experimental): An AI software device (AEYE-DS) to be used as a diagnostic tool to assist primary care clinicians in screening for diabetic retinopathy using digital funduscopic images. The device automatically detects more than mild diabetic retinopathy (mtmDR) in adults diagnosed with diabetes who have not been previously diagnosed with diabetic retinopathy.
  Interventions: Device: AEYE Software Device

INTERVENTIONS:
Device: AEYE Software Device — Eligible participants will undergo the following procedures:
  * Photographic imaging of each eye using a funduscopy camera device. Images obtained will be sent to the AEYE-DS software for analysis.
  * Additional photographic and Optical Coherence Tomography (OCT) images will be obtained using a second funduscopy/OCT camera device. Images obtained will be sent to a professional reading center for analysis.
  * All study subjects will have their pupils dilated using dilation drops.

SUMMARY:
AEYE-DS is a software device developed to increase compliance with diabetic retinopathy screening by automatically detecting more-than-mild diabetic retinopathy from digital fundus images using Artificial Intelligence (AI)-based software. This study has been designed to validate the safety and efficacy of the device at primary care and other point of care sites.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22
* Male or female
* Documented diagnosis of diabetes mellitus, meeting the criteria established by the American Diabetes Association (ADA) and World Health Organization (WHO).
* Understand the study and volunteer to sign the informed consent

Exclusion Criteria:

* Uncorrectable vision loss (e.g., with the use of eyeglasses), blurred vision, or floaters.
* Diagnosed with macular edema, severe non-proliferative retinopathy, proliferative retinopathy, radiation retinopathy, or retinal vein occlusion.
* History of laser treatment of the retina or injections into either eye, or any history of retinal surgery.
* Currently participating in another investigational eye study and actively receiving investigational product for Diabetic Retinopathy (DR) or Diabetic Macular Edema (DME).
* Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure or glycemic control, microphthalmia or previous enucleation).
* Participant is contraindicated for imaging by fundus imaging systems used in the study:

  1. Participant is hypersensitive to light
  2. Participant recently underwent photodynamic therapy (PDT)
  3. Participant is taking medication that causes photosensitivity
  4. Participant has a history of angle-closure glaucoma or narrow anterior chamber angles

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-12-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Eye Care Institute, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AEYE Software Device: An AI software device (AEYE-DS) to be used as a diagnostic tool to assist primary care clinicians in screening for diabetic retinopathy using digital funduscopic images. The device automatically detects more than mild diabetic retinopathy (mtmDR) in adults diagnosed with diabetes who have not been previously diagnosed with diabetic retinopathy.
  AEYE Software Device: Eligible participants will undergo the following procedures:
  * Photographic imaging of each eye using a funduscopy camera device. Images obtained will be sent to the AEYE-DS software for analysis.
  * Additional photographic and OCT images will be obtained using a second funduscopy/OCT camera device. Images obtained will be sent to a professional reading center for analysis.
  * All study subjects will have their pupils dilated using dilation drops.
Period: Overall Study
Arm/Group | AEYE Software Device
Started | 531 (screened and enrolled)
Analyzable | 468
Completed | 462 (participants included in statistical analysis with fully analyzable data with valid ground truth (based on worst eye analysis) and AEYE-DS results output per participant.)
Not Completed | 69

BASELINE CHARACTERISTICS:
Population: Full Analysis (FA) Set - includes all eligible patients who were enrolled in and completed the study with analyzable data
Arm/Group | AEYE Software Device
Number analyzed (Participants) | 468
Age, Continuous [Mean (Full Range); unit: years] | 55 [21 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246
  Male | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 138
  Not Hispanic or Latino | 329
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 132
  White | 323
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 440
  Israel | 28

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity, Based on Two Macula-centered Images (One Image From Each Eye of the Patient)
Description: Sensitivity and specificity of the AEYE-DS device to detect mtmDR on digital funduscopic images, acquired by the Topcon NW400 fundoscopy device, based on two macula-centered images (one image from each eye of the patient). Sensitivity and specificity were calculated by comparing the output results of the AEYE-DS device to the ground truth (diagnostic determination by an independent, blinded panel of expert ophthalmologists at a reading center). The worst of two eyes was compared with the AEYE-DS output at the participant level.
Time Frame: 1 day
Population: Completed subjects with valid ground truth and AEYE-DS results
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AEYE Software Device
Number analyzed (Participants) | 462
percentage of participants
  Sensitivity | 92.98 [83.3 to 97.24]
  Specificity | 91.36 [88.22 to 93.72]

2. Secondary Outcome: Sensitivity and Specificity, Based on Four Images (One Macula Centered Image and One Optic Disc Centered Image Per Eye)
Description: Sensitivity and specificity of the AEYE-DS device to detect mtmDR from digital funduscopic images, acquired by the Topcon NW400 fundoscopy device, based on four images (one macula centered image and one optic disc centered image per eye). Sensitivity and specificity were calculated by comparing the output results of the AEYE-DS device to the ground truth (diagnostic determination by an independent, blinded panel of expert ophthalmologists at a reading center). The worst of two eyes was compared with the AEYE-DS output at the participant level.
Time Frame: 1 day
Population: completed subjects with valid ground truth and AEYE-DS results
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AEYE Software Device
Number analyzed (Participants) | 462
percentage of participants
  Sensitivity | 94.74 [85.63 to 98.19]
  Specificity | 88.64 [85.18 to 91.38]

3. Secondary Outcome: Imageability, Based on Two Macula-centered Images (One Image From Each Eye of the Patient)
Description: To assess the imageability of AEYE-DS, defined as the percentage of participants with a diagnostic output (positive for more than mild DR or negative for more than mild DR) from the AEYE-DS device. Participants with no diagnostic output (i.e., AEYE-DS output of "Insufficient Quality") lowers the imageability of the AEYE-DS.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AEYE Software Device
Number analyzed (Participants) | 462
percentage of participants | 99.1 [97.8 to 99.7]

4. Secondary Outcome: Imageability, Based on Four Images (One Macula Centered Image and One Optic Disc Centered Image Per Eye)
Description: as for outcome 3
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AEYE Software Device
Number analyzed (Participants) | 462
percentage of participants | 99.1 [97.8 to 99.7]

ADVERSE EVENTS:
Time Frame: Since this study was non-interventional with regards to the AEYE-DS device (i.e., it did not come in contact with the study participants) and all interventions were conventional screening exams with FDA-cleared devices used to obtain all of the ophthalmic examinations, information about adverse events was not collected. No safety assessments were necessary.
Description: Since this study was non-interventional with regards to the AEYE-DS device (i.e., it did not come in contact with the study participants) and all interventions were conventional screening exams with FDA-cleared devices used to obtain all of the ophthalmic examinations, information about adverse events was not collected. No safety assessments were necessary.
Arm/Group | AEYE Software Device
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04612868/Prot_SAP_000.pdf